CLINICAL TRIAL: NCT01681303
Title: Effect of An Oral Absorbent AST-120 in Late-stage Chronic Kidney Disease (CKD) Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, iwenwu, Attending Physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IWW-0004; 98-794A3 (Other Grant/Funding Number: Conmed)
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Kidney Disease; AST-120
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — AST 120

ARMS (2):
- AST-120 group (Experimental): Administration of AST-120
  Interventions: Drug: AST-120
- 2 (No Intervention)

INTERVENTIONS:
Drug: AST-120
  Arms: AST-120 group

SUMMARY:
Recent research work has directed especial attention toward a distinct group of uremic retension molecules, called "protein-bound uremic toxins". The prototypes of this group of uremic toxins are indoxyl sulfate and p-cresol. These uremic toxins can promote production of free radical and impair antioxidant system and exerts direct toxicity on different cells and organs, including mesangial, tubular, endothelial cell and osteoblasts. Accumulation of these protein bound uremic toxins results in glomerular sclerosis and interstitial fibrosis of kidneys of uremic rats and confer skeletal resistance to parthyroid hormone in uremic patients. In hemodialysis, high serum p-cresol level is associated with higher cardiovascular mortality.

AST-120 (Kremezin) is a carbonated oral absorbent extensively used in Japan and Korea. It has superior adsorption ability for certain small-molecular weight organic compounds known to accumulate in patients with CKD. In uremic rats and CKD patients, oral administration of AST-120 decreased the elevated pretreatment levels of serum indoxyl sulfate. In Japan, it was reported that AST-120 suppressed the increase in serum creatinine levels, prevented proteinuria, improved uremic symptoms, and, consequently, led to the postponement of dialysis therapy.

Value of AST-120 on the outcome of late-stage CKD patients is still unknown. We hypothesized AST-120 through reduction of level of indoxyl sulfate and p-cresol can improved the morbidity- mortality of CKD patients.

The principal aim of this prospective cohort study is to investigate the effectiveness of AST-120 in incidence of dialysis and mortality of late-stage CKD patients. Determination of this relationship can help to establish new therapeutic strategy in the treatment of late-stage CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* adults aged > 18 year-old or < 85 year-old
* eGFR or CCR < 60 ml/min
* hemoglobin < 10 g/dL, ESA-naïve, had adequate iron storage (serum ferritin > 200 ng/dL and transferrin saturation > 20%)
* no spontaneous renal improvement or progression in past 3 months.

Exclusion Criteria:

* renal transplant recipients, liver cirrhosis, bone marrow disorder
* blood pressure > 170/80 mmHg in 3 occasions
* recent cardiovascular disease (Coronary artery disease, myocardial ischemia, cerebrovascular disease or peripheral artery disease) or gastrointestinal bleeding in past 3 months
* acute tubular necrosis in the past 3 months
* unwilling to participate in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
renal function change | 1 year

SECONDARY OUTCOMES:
anemia | 1 year

OTHER OUTCOMES:
lipid profile and uric acid | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: I-Wen Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Nephrology, Chang Gung Memorial Hospital, Keelung, Taiwan